CLINICAL TRIAL: NCT00990912
Title: A Study to Document Long-term Safety and Continued Benefit of Irinotecan and Carboplatin or Irinotecan in Subjects 1 - 21 Years of Age With Refractory Solid Tumors Who Have Experienced Clinical Benefit Following a Minimum of 6 Cycles of Therapy on BMS Protocol CA124-001 or BMS Protocol CA124-002
Brief Title: A Study to Document Long-Term Safety and Continued Benefit of Irinotecan and Carboplatin or Irinotecan in Subjects With Refractory Solid Tumors (Rollover Study -001, -002)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA124-003
Record Dates: First submitted 2009-10-05; First posted 2009-10-07 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2009-10

CONDITIONS: Pediatric Solid Tumors
MeSH Terms: interventions — Carboplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Carboplatin (Experimental)
  Interventions: Drug: Carboplatin
- Irinotecan (12 (9) mg/m²/day) (Experimental)
  Interventions: Drug: Irinotecan
- Irinotecan (10 (10) mg/m²/day (Active Comparator)
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Carboplatin — IV, Infusion, AUC2 mg/ml.min, Once every 21 days, until progression or unacceptable toxicity
  Other Names: Paraplatin; BMY-26575
  Arms: Carboplatin
Drug: Irinotecan — IV, Infusion, 12 (9) mg/m²/day, Once daily x 10 days, every 21 days, until progression or unacceptable toxicity
  Other Names: Camptosar; Campto
  Arms: Irinotecan (12 (9) mg/m²/day)
Drug: Irinotecan — IV, Infusion, 10 (18) mg/m²/day, Once daily x 10 days, every 21 days, until progression or unacceptable toxicity
  Other Names: Camptosar; Campto
  Arms: Irinotecan (10 (10) mg/m²/day

SUMMARY:
The purpose of this study is to determine the long term safety of patients with refractory solid tumors who have experienced clinical benefit after at least 6 cycles of treatment in BMS Protocol CA124-001 or CA124-002.

ELIGIBILITY:
Inclusion Criteria:

* Completion of at least 6 cycles of therapy on BMS clinical protocol CA124-001 or CA124-002 and who continue to derive clinical benefit and are not experiencing intolerable toxicity from the therapy
* Karnofsky score of at least 50 for subjects > 10 years of age; Lansky play scale of at least 50 for children 10 years of age and younger
* Recovery to baseline or Grade 1 from toxicities (except alopecia or asthenia) resulting from previous therapies
* Males and females, ages 1 - 21 years of age at the time of consent into CA124-001 or CA124-002

Exclusion Criteria:

* A serious uncontrolled medical disorder that in the opinion of the Investigator would impair the ability of the subject to receive protocol therapy
* Requirement to receive concurrent chemotherapy, immunotherapy, radiotherapy, or any other investigational drug while on study
* Inadequate bone marrow and renal function
* Concurrent receipt of Dilantin®(phenytoin), phenobarbital, primidone, Tegretol®(carbamazepine), Depacon®, Depakene®, Depakote®, and Deproic®(valproic acid)

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2004-01; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Assessment of safety and tolerability | 22 months

SECONDARY OUTCOMES:
Assessment of duration of clinical benefit per CT or MRI, steroid use and neuropathy assessment | Every other cycle for 22 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb